CLINICAL TRIAL: NCT03640286
Title: Clinical Investigation Protocol for the Demonstration of Safety and Efficacy of VeSTAL Weight Loss Device in Human Subjects. Randomized Study of VeSTAL in Patients Who Are Overweight
Brief Title: Vestibular Stimulation to Trigger Adipose Loss (VeSTAL) Clinical Trial
Acronym: VeSTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University of California, San Diego (Other); University of Ulster (Other); Exploristics (Unknown); Compliance Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243973
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: Overweight; Metabolic syndrome; Weight loss; Diet; Atherogenic index; Prediabetes
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome; Weight Loss; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VeSTAL - active device (Active Comparator): The VeSTAL device utilizes a technology called galvanic vestibular stimulation (GVS) (sometimes termed vestibular nerve stimulation (VeNS)). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day.
  Interventions: Device: VeSTAL
- Sham device (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. However, it does not deliver vestibular stimulation to users. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 1 hour per day.
  Interventions: Device: VeSTAL

INTERVENTIONS:
Device: VeSTAL — The aim of this study is to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation in combination with a lifestyle modification program, as a method of reducing excess body weight and body fat, as compared to a sham device in combination with the same lifestyle modification program.

SUMMARY:
A randomized, double blind sham controlled clinical trial to evaluate the efficacy of vestibular nerve stimulation (VeNS), combined with a lifestyle modification program, compared to a sham control and a lifestyle modification program as a means of reducing excess body weight and body fat.

The purpose of this investigation device study is to collect data to support regulatory submissions, primarily in the United States of America (USA), but it may also be used to support submissions in other regions, including the European Union (EU).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation (VeNS), together with a lifestyle modification program, as a method of reducing excess body weight and body fat, as compared to a sham control with both study arms incorporating a lifestyle modification program.

* Allocation: Randomized
* Endpoint classification: Efficacy Study
* Intervention Model: Parallel Assignment in 1:1 active to control allocation
* The aim of the study is to recruit a total (i.e. across all 4 sites) of 200 participants that pass the screening process and are randomized into the treatment protocols. With a dropout allowance of 10% this should generate a minimum of 90 active treatment and 90 control subjects.
* Masking: Double Blind (Subject, Nursing staff, Dietician, Co-coordinators, Outcomes Assessor and any other study staff who have contact with the subject)
* Data from all sites will be collated at the end of the studies and analysis will be performed on one data set.

This protocol governs the activities at both the USA and NI/UK clinical sites.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Body mass index BMI ≥ 27 kg/m2.
3. Males or Females. Note females of child-bearing potential must have a negative urine pregnancy test at screen and also just before each DXA scan. (As DXA involves a small dose of ionizing radiation). They should agree to follow a physician-approved contraceptive regimen for the duration of the study period (other than DMPA injections as this causes weight gain).
4. 22-80 years of age inclusive on starting the study. (In order to comply with FDA guidance: https://www.fda.gov/MedicalDevices/DeviceRegulationandGuidance/GuidanceDocuments/ucm089740.htm#s6)
5. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with: trying to use the device on a daily basis; the hypocaloric diet weight loss program; and this provided weight loss support and mentoring.
6. Agreement not to use of prescription, or over-the-counter, weight loss preparations for the duration of the trial.
7. Agreement not to start smoking tobacco or marijuana

Exclusion Criteria:

1. History of vestibular dysfunction or other inner ear disease as indicated by the screening questions.
2. History of bariatric surgery, or gastric resection.
3. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
4. History of weight loss device implantation (e.g. VBloc Maestro or Abiliti).
5. Use of a non-invasive weight loss device (e.g. Modius)
6. Hypothyroidism requiring current treatment with levothyroxine (e.g. Levo-T, Synthroid, Thyroxine) (Other thyroid disorder patients on stable treatment for at least 3 months are acceptable).
7. Other endocrinological causes of weight gain (e.g. Cushing's disease, Cushing's syndrome or acromegaly)
8. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working).
9. Diagnosis of cirrhosis, chronic pancreatitis, or liver, kidney or heart failure.
10. Treatment with prescription weight-loss drug therapy in the 6 months before starting the study.
11. Tobacco smoking (including vaping) in the six months prior to starting and for the duration of the study.
12. Use of marijuana (smoking, vaping or in edible form) more than twice a month on average.
13. Known genetic cause of obesity (e.g., Prader-Willi Syndrome).
14. Body weight change of more than 20% in either direction within the previous year.
15. Physician-prescribed diet, and/ or current, active member of an organized weight loss program.
16. Diabetes mellitus (Types 1 & 2).
17. Diagnosis of epilepsy or use of anti-epileptic medication within six months of starting the study (e.g. for the treatment of peripheral neuropathy)
18. Chronic (more than a month of daily use) treatment with opioid analgesic drugs within the last 6 months.
19. Regular use (more than twice a month) of anti-histamine medication within the last 6 months.
20. Use of oral or intravenous corticosteroid medication within 6 months of starting the study.
21. Use of the beta-blockers atenolol, metoprolol or propranolol within 3 months of starting the study.
22. Current alterations in treatment regimens of anti-depressant medication for whatever reason (including tricyclic antidepressants) (Note: stable treatment regimen for prior 6 months acceptable).
23. An active diagnosis of cancer.
24. A myocardial infarction within the preceding year.
25. A history of stroke or severe head injury (as defined by a head injury that required craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).
26. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
27. Psychiatric disorders (including untreated severe depression, schizophrenia, substance abuse, eating disorder etc.)
28. Current participant in another weight loss study or other clinical trial.
29. Have a family member who is currently participating or is planning to participate in this study.
30. Weight over 350 pounds at UU, TDE and CTRI site (as this is the weight limit of the DXA scanner) or a weight over 500 pounds at the EPARC site (as this is the weight limit of the DXA scanner)
31. Pregnancy The decision to exclude participants with type 2 diabetes mellitus was made after reading the FDA's draft guidance (see: http://www.fda.gov/downloads/Drugs/.../Guidances/ucm071612.pdf). This notes that, "[c]compared with nondiabetic patients, overweight and obese patients with type 2 diabetes often respond less favorably to weight-management products and may face unique safety issues such as risk for sulfonylurea-induced hypoglycemia following weight loss (if the dose of sulfonylurea is not appropriately lowered or the drug discontinued)." The FDA then go on to advise "examining the efficacy and safety of weight-management products in trials dedicated to patients with type 2 diabetes." On the basis of this advice we made the decision to exclude patients with type 2 diabetes. This is an important patient group of course, and our intention is to investigate type 2 diabetics in due course.

If a subject is found to possibly have type 2 diabetes during the initial screening, then they will be excluded and asked to notify their primary care physician. However, if a subject passes the initial screening but a suspicion of this diagnosis arises during one of the study tests, then the subject will be asked to notify their primary care physician, though they will still be allowed to complete the study.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Viirre, MD PhD, Principal Investigator — UC San Diego
Locations (4):
- United States (3):
  - UC San Diego, Exercise and Physical Activity Resource Center, La Jolla, California
  - University of California San Diego, Altman Clinical & Translational Research Institute,, La Jolla, California
  - Texas Diabetes and Endocrinology, Austin, Texas
- Univeristy of Ulster, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be transferred in an encrypted PDF format. Trial staff will be given direction on how to share the trial data and given access to one specific section of a controlled cloud service which is controlled via role based access. Once they have authenticated with the service and the service verifies that they have the correct role to access the system they will be directed to a single webpage within the application where they will be able to upload the encrypted PDF. This PDF is generated on the fly and is therefore not stored in another location that could become compromised. Generating the PDF on the fly means that the source data is extracted from the database, processed and delivered in the context of a single request. These data will be transferred for each subject when they complete participation in the study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VeSTAL - Active Device | Sham Device
Started | 117 | 124
Completed | 91 | 89
Not Completed | 26 | 35
Not completed — Adverse Event | 6 | 6
Not completed — Lost to Follow-up | 3 | 6
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Non-compliance | 4 | 10
Not completed — Medication change | 1 | 0
Not completed — Other | 1 | 2
Not completed — Joined another lifestyle program | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VeSTAL - Active Device | Sham Device | Total
Number analyzed (Participants) | 117 | 124 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.3) | 47.2 (10.8) | 46.3 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 99 | 198
  Male | 18 | 25 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 6 | 9 | 15
  White | 94 | 95 | 189
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 71 | 76 | 147
  United Kingdom | 46 | 48 | 94
Weight [Mean (Standard Deviation); unit: Kg] | 99.60 (20.07) | 99.86 (20.37) | 99.73 (20.18)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 36.94 (6.65) | 35.81 (5.76) | 36.36 (6.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of Weight From Baseline
Description: The mean percentage weight loss achieved by the Vestal active device in comparison to the sham device
Time Frame: From baseline to 6 months
Population: Unadjusted Intention to treat analysis
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 91 | 90
Percentage change from baseline | -2.46 (4.766) | -1.97 (4.971)

2. Primary Outcome: Categorical: Proportion of Participants Who Lose 5% Total Body Weight
Description: The proportion of participants who lose 5% total body weight or more in the active Vestal group is at least 50%, independent of the sham control
Time Frame: 6 months
Population: Unadjusted Intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 117 | 124
Participants | 25 | 25

3. Secondary Outcome: Mean Percent Loss of Baseline Visceral Adipose Tissue
Description: The difference in mean percent loss of baseline visceral adipose tissue in the active versus placebo treated groups. (As measured by a whole body DXA scan).
Time Frame: % change in VAT mass at 6 months
Population: Unadjusted Intention to treat
Measure: Mean (Standard Deviation); unit: % change in VAT mass at 6 months
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 54 | 58
% change in VAT mass at 6 months | -10.316 (12.4607) | -4.731 (14.6057)

4. Secondary Outcome: Percentage Fat Loss
Description: Percentage fat loss from baseline. (As measured by means of a whole body DXA scan).
Time Frame: Percentage change from baseline to 6 months
Population: Unadjusted Intention to Treat
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 60 | 58
Percentage change | -5.268 (8.1254) | -3.638 (9.1772)

5. Secondary Outcome: Difference in Lean Muscle Mass in the Active Versus Placebo Treated Group
Description: Difference in lean muscle mass (in kilograms) in the active versus placebo treated group. (As measured by the whole body DXA scan).
Time Frame: Absolute change at 3 months and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 9 | 8
Kg
  3 months | -0.107 (2.1676) | 0.990 (1.3227)
  6 months | -0.169 (1.9577) | -0.078 (1.8110)

6. Secondary Outcome: Atherogenic Index
Description: The Atherogenic Index is calculated using the lipid profile by determining the ratio of Total Cholesterol (TC) to High-Density Lipoprotein (HDL) cholesterol.
  If the ratio has been transformed (e.g., natural log-transformed or log10), this will be explicitly stated in the analysis, and the Unit of Measure will reflect this transformation as "log(ratio)" or "ln(ratio)" accordingly.
Time Frame: Absolute change from baseline to 6 months
Population: Unadjusted Intention to Treat
Measure: Mean (Standard Deviation); unit: Atherogenic Index
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 55 | 55
Atherogenic Index | -0.10 (0.660) | -0.27 (0.454)

7. Secondary Outcome: Systemic Inflammation
Description: Systemic inflammation is assessed using high-sensitivity C-reactive protein (hs-CRP) levels, measured in milligrams per liter (mg/L). This outcome measure represents the percentage change in hs-CRP levels from baseline to 6 months.
  Higher or lower percentage changes indicate increases or decreases in systemic inflammation, respectively. Values are reported as the mean percentage change with standard deviation (SD) for each group.
Time Frame: Percentage change from baseline to 6 months
Population: Unadjusted Intention to Treat
Measure: Mean (Standard Deviation); unit: % change mg/ml
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 57 | 56
% change mg/ml | -0.51 (5.645) | -0.31 (1.845)

8. Secondary Outcome: Total Energy Intake (kcal)
Description: Total Energy intake (kcal) as assessed by two-day 24 hour dietary recall.
Time Frame: Change from baseline to 6 months
Population: Unadjusted
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 82 | 85
kcal | -241.56 (703.820) | -180.39 (1114.909)

9. Secondary Outcome: Quality of Life Ratings
Description: Quality of life was assessed using the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) questionnaire, a validated self-report measure designed to assess obesity-specific quality of life in adults. Scores range from 0 to 100, with higher scores indicating better quality of life.
  The outcome measure reflects the absolute change in IWQOL-Lite total scores from baseline to 6 months (i.e., IWQOL-Lite score at 6 months minus IWQOL-Lite score at baseline). Results are reported as the mean absolute change with standard deviation for each study arm.
Time Frame: Absolute change from baseline to 6 months
Population: Adjusted Intention to Treat
Measure: Mean (Standard Deviation); unit: IWQoL Total Score
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 88 | 89
IWQoL Total Score | 7.71 (12.193) | 9.08 (14.022)

10. Other Pre Specified Outcome: Baseline Truncal Body Fat
Description: This outcome measure assesses the amount of body fat located in the trunk or torso region at baseline. Truncal body fat includes both visceral and subcutaneous fat around the abdomen, chest, and back. It is typically measured using a whole-body DXA scan, which provides an accurate assessment of fat distribution. The baseline value is recorded before any intervention or treatment to serve as a reference point for evaluating changes in truncal body fat over the course of the study.
Time Frame: Baseline
Population: ITT
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 117 | 124
Kg | 25.209 (8.4520) | 24.393 (7.4186)

11. Other Pre Specified Outcome: 6 Month Truncal Body Fat
Description: as for outcome 10
Time Frame: 6 Month
Population: ITT
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 10 | 8
Kg | 19.082 (4.1085) | 20.008 (4.5043)

12. Other Pre Specified Outcome: Difference in Bone Mineral Content
Description: Bone mineral content (BMC) was measured to assess changes in bone health. The outcome reflects the absolute change in BMC from baseline to 6 months (i.e., BMC at 6 months minus BMC at baseline). Results are reported as the mean absolute change with standard deviation (SD) for each study arm.
  The Unit of Measure is BMC (kg), consistent with the reported data. Higher values indicate greater BMC, while lower or negative values indicate reductions in BMC over time.
Time Frame: Absolute change from baseline to 6 months
Population: Unadjusted Intention to Treat
Measure: Mean (Standard Deviation); unit: BMC (kg)
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 60 | 58
BMC (kg) | 0.003 (0.0645) | -0.001 (0.0504)

13. Other Pre Specified Outcome: Fasting Glucose Change From Baseline
Description: Fasting glucose in mg/dL
Time Frame: Change from Baseline to 6 months
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 55 | 56
mg/dl | 0.798 (10.9941) | 0.164 (6.8325)

14. Other Pre Specified Outcome: Glycated Hemoglobin
Description: This outcome measures the change in glycated hemoglobin (HbA1c) levels, reported as a percentage (%), from baseline to 6 months. HbA1c is a biomarker that reflects average blood glucose levels over the past 2-3 months and is commonly used to assess long-term glucose control. A reduction in HbA1c indicates improved blood sugar management. The change is calculated by subtracting the baseline value from the value at 6 months.
Time Frame: Change from baseline to 6 months Change from baseline to 6 months Change from baseline to 6 months
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 56 | 56
percentage of HbA1c | -0.148 (0.8657) | -0.004 (0.2166)

15. Other Pre Specified Outcome: Blood Pressure
Description: This outcome measures the change in diastolic blood pressure (measured in mmHg). Diastolic blood pressure was assessed using standard clinical methods at each time point.
Time Frame: Baseline
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 119
mmHg | 85.4 (11.07) | 82.0 (10.10)

16. Other Pre Specified Outcome: Blood Pressure
Description: as for outcome 15
Time Frame: 6 Months
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 59 | 58
mmHg | 85.6 (11.46) | 81.3 (8.89)

17. Other Pre Specified Outcome: Heart Rate
Description: Heart rate in beats per minute
Time Frame: Baseline and 6 months
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 119
bpm
  Baseline | 70.8 (9.99) | 69.6 (10.14)
  6 months: number analyzed (Participants) | 59 | 58
  6 months | 71.1 (10.29) | 68.6 (10.66)

18. Other Pre Specified Outcome: Hip-waist Ratio
Description: Hip-waist ratio
Time Frame: 6 months
Population: Data not analysed
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: BMI in kg/m^2
Time Frame: Baseline and 6 months
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 116 | 122
kg/m^2
  Baseline | 36.9 (6.68) | 35.9 (5.78)
  6 months: number analyzed (Participants) | 91 | 90
  6 months | 36.6 (6.94) | 34.8 (6.25)

20. Other Pre Specified Outcome: Concomitant Medication: Cardiovascular Adjustments and Weight Gain Causality
Description: This outcome measure tracks the use of concomitant medications during the study, focusing on adjustments in cardiovascular medications and the presence of medications known to influence weight. For cardiovascular medications, data include any increases, decreases, or no changes in medication use, as well as instances where information is not applicable (N/A). The assessment also includes the categorization of medications known to cause weight gain or weight loss, reporting the number of participants using such medications. This allows for an understanding of how changes in cardiovascular treatments and the use of weight-altering medications may interact with study outcomes.
Time Frame: Baseline, Month 3, Month 6 (or other specified time points)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 117 | 124
Participants
  Increase in cardiovascular medication | 2 | 4
  Decrease in cardiovascular medication | 1 | 3
  No change in cardiovascular medication | 24 | 28
  N/A | 1 | 0
  Not reported | 89 | 89

21. Other Pre Specified Outcome: Concomitant Medication: Cardiovascular Adjustments and Weight Gain Causality
Description: as for outcome 20
Time Frame: Baseline, Month 3, Month 6 (or other specified time points)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 117 | 124
Participants
  Medication knwon ro cause weight gain | 34 | 42
  Medication known to cause weight loss | 23 | 29
  Not reported | 60 | 53

22. Other Pre Specified Outcome: Dose Response Analysis
Description: It is likely that some subjects will use their device more than other. Usage data will be available from the devices permitting a dose response analysis, which will done be in an intention to treat manner.
  Treatment Compliance =(Number of weeks with over 5 hours of total usage / Number weeks of device usage)*100 High Treatment Compliance = Treatment Compliance >75% Medium Treatment Compliance = Treatment Compliance >=55% and <=75% Low Treatment Compliance = Treatment Compliance <55%
Time Frame: Percentage Weight Loss from Baseline, by Treatment and Treatment Compliance at 3 months and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: % weight loss
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 117 | 124
% weight loss
  Month 3 High: number analyzed (Participants) | 22 | 22
  Month 3 High | -2.60 (3.105) | -3.51 (3.951)
  Month 3 Medium: number analyzed (Participants) | 13 | 15
  Month 3 Medium | -2.48 (2.825) | -1.38 (3.276)
  Month 3 Low: number analyzed (Participants) | 63 | 57
  Month 3 Low | -1.79 (3.060) | -0.84 (2.939)
  Month 6 High: number analyzed (Participants) | 23 | 23
  Month 6 High | -4.26 (4.070) | -4.73 (5.223)
  Month 6 Medium: number analyzed (Participants) | 11 | 14
  Month 6 Medium | -3.64 (3.490) | -1.24 (5.407)
  Month 6 Low: number analyzed (Participants) | 57 | 53
  Month 6 Low | -1.46 (4.320) | -1.00 (4.073)

23. Other Pre Specified Outcome: Hearing Loss Assessment
Description: Hearing Loss (Judged to be abnormal, normal or missing by examining clinician by audiometry results).
Time Frame: Baseline and 6 months
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 116 | 122
Participants
  Baseline: Abnormal | 7 | 3
  Baseline: Normal | 109 | 119
  Baseline: Missing | 0 | 0
  Month 6: Abnormal | 6 | 3
  Month 6: Normal | 73 | 77
  Month 6: Missing | 37 | 42

24. Other Pre Specified Outcome: Food Frequency Questionnaire
Description: This outcome measure evaluates nutrient intake based on responses from the Food Frequency Questionnaire (FFQ). The FFQ assesses the frequency of consumption of various food items, allowing for an estimation of intake for several nutrients, including energy (kcal), carbohydrates (g), free sugars (g), total sugars (g), starch (g), fat (g), saturated fat (g), protein (g), fiber (g), and alcohol (g). Participants report their typical consumption of foods and beverages, which is then used to estimate their average intake of these nutrients over a specified period. The data are reported in grams or kilocalories, as appropriate for each nutrient, and can be used to evaluate dietary patterns and nutrient consumption changes throughout the study.
Time Frame: Baseline
Population: ITT
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 109 | 114
grams
  Carbohydrate | 230.95 (128.239) | 234.69 (171.041)
  Free sugars | 62.97 (53.947) | 65.86 (80.208)
  Sugars | 122.17 (79.046) | 130.20 (104.795)
  Starch | 99.92 (61.226) | 96.03 (67.388)
  Fat | 117.40 (58.807) | 113.19 (70.277)
  Saturated Fat | 46.55 (26.980) | 43.76 (32.643)
  Protein | 130.21 (46.945) | 124.81 (61.433)
  Fibre | 28.48 (22.071) | 29.69 (15.287)
  Alcohol | 5.3 (8.302) | 5.41 (9.922)

25. Other Pre Specified Outcome: Fat Intake
Description: Fat intake as assessed by 24 hour dietary recall.
Time Frame: Baseline, 3-months and 6-months
Population: ITT
Measure: Mean (Standard Deviation); unit: Fat (g)
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 122
Fat (g)
  Baseline | 78.73 (38.935) | 78.51 (37.884)
  Month 3: number analyzed (Participants) | 93 | 89
  Month 3 | 66.15 (25.570) | 67.08 (32.377)
  Month 6: number analyzed (Participants) | 83 | 85
  Month 6 | 71.89 (28.724) | 72.87 (68.834)

26. Other Pre Specified Outcome: Carbohydrate; Starchy Carbohydrates, Sugars, and Free Sugars
Description: Carbohydrate; starchy carbohydrates, sugars, and free sugars (grams) as assessed by 24 hour dietary recall
Time Frame: Baseline, 3-months and 6-months
Population: ITT
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 122
grams
  Baseline | 191.68 (79.983) | 188.01 (84.253)
  Month 3: number analyzed (Participants) | 93 | 89
  Month 3 | 170.88 (64.303) | 165.94 (66.797)
  Month 6: number analyzed (Participants) | 83 | 85
  Month 6 | 158.55 (69.894) | 178.29 (159.162)

27. Other Pre Specified Outcome: Fiber
Description: Fiber (grams) as assessed by 24 hour dietary recall and Food Frequency Questionnaire
Time Frame: Baseline, 3-months and 6-months
Population: ITT
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 122
grams
  Baseline | 19.31 (7.831) | 19.54 (8.989)
  Month 3: number analyzed (Participants) | 93 | 89
  Month 3 | 19.79 (7.938) | 18.61 (9.378)
  Month 6: number analyzed (Participants) | 83 | 85
  Month 6 | 18.25 (6.570) | 18.62 (9.227)

28. Other Pre Specified Outcome: Alcohol
Description: This outcome measure assesses alcohol consumption (in grams) based on a two-day, 24-hour dietary recall. Participants were asked to recall their alcohol intake for two separate 24-hour periods, providing a comprehensive estimate of their usual consumption. The data is presented for baseline, 3-month, and 6-month time points, with values reported as the mean and standard deviation (SD).
Time Frame: Baseline, 3-month, and 6-month
Population: ITT
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 37 | 40
grams
  Baseline | 23.67 (17.900) | 26.38 (20.501)
  Month 3: number analyzed (Participants) | 25 | 28
  Month 3 | 22.45 (17.948) | 16.63 (11.682)
  Month 6: number analyzed (Participants) | 31 | 28
  Month 6 | 25.02 (23.928) | 21.63 (20.519)

29. Other Pre Specified Outcome: Healthy Eating Index
Description: Nutrient intakes assessment from two-day 24-hour recall. Score out of 100 with a higher score reflecting a better quality of diet.
Time Frame: 6 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Total Physical Activity in MET-hours Per Week
Description: Total Physical Activity averaged over the past year in MET-hours per week as assessed by the Modifiable Activity Questionnaire
Time Frame: Baseline and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: MWET-hours/Week
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 114 | 119
MWET-hours/Week
  Baseline | 57.19 (83.990) | 43.17 (58.502)
  Month 6: number analyzed (Participants) | 87 | 88
  Month 6 | 41.19 (53.354) | 41.85 (57.977)

31. Other Pre Specified Outcome: Saturated Fat Intake
Description: Saturated fat intake as assessed by 24 hour dietary recall.
Time Frame: Baseline, 3-months and 6-months
Population: ITT
Measure: Mean (Standard Deviation); unit: Saturated Fat (g)
Arm/Group | VeSTAL - Active Device | Sham Device
Number analyzed (Participants) | 115 | 122
Saturated Fat (g)
  Baseline | 26.11 (14.820) | 27.16 (15.163)
  Month 3: number analyzed (Participants) | 93 | 89
  Month 3 | 22.33 (12.765) | 22.23 (12.678)
  Month 6: number analyzed (Participants) | 83 | 85
  Month 6 | 24.73 (12.761) | 25.97 (28.760)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | VeSTAL - Active Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/122
Other Adverse Events (participants affected / at risk) | 52/116 | 56/122
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VeSTAL - Active Device (N=116) | Sham Device (N=122)
Dizziness (Nervous system disorders) | 24 | 37
Fatigue (General disorders) | 18 | 19
Headache (Nervous system disorders) | 18 | 12
Ear Pain (Ear and labyrinth disorders) | 13 | 11
Mild Tinnitus (Ear and labyrinth disorders) | 18 | 4
Skin Irritation (Skin and subcutaneous tissue disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03640286/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03640286/SAP_001.pdf